CLINICAL TRIAL: NCT01992263
Title: A Trial of Vitamin D Supplementation Among Tuberculosis Patients in South India
Brief Title: Vitamin D Supplementation and TB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cornell University (Other)
Collaborators: Arogyavaram Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB #: 1304003801
Record Dates: First submitted 2013-11-01; First posted 2013-11-25 (Estimated); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Tuberculosis; Vitamin D; Immunity
Keywords: tuberculosis; vitamin D; immunity
MeSH Terms: conditions — Tuberculosis | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vitamin D (600 IU) (Experimental)
  Interventions: Dietary Supplement: Vitamin D (600 IU)
- Vitamin D (2000 IU) (Experimental)
  Interventions: Dietary Supplement: Vitamin D (2000 IU)
- Vitamin D (4000 IU) (Experimental)
  Interventions: Dietary Supplement: Vitamin D (4000 IU)
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D (600 IU) — Daily oral dose for 12 months
  Arms: Vitamin D (600 IU)
Dietary Supplement: Vitamin D (2000 IU) — Daily oral dose for 12 months
  Arms: Vitamin D (2000 IU)
Dietary Supplement: Vitamin D (4000 IU) — Daily oral dose for 12 months
  Arms: Vitamin D (4000 IU)
Other: Placebo — Daily oral dose for 12 months
  Arms: Placebo

SUMMARY:
The goal of this study is to understand the effects of vitamin D supplementation on immunological outcomes among patients with tuberculosis.

DETAILED DESCRIPTION:
In this randomized trial, the investigators will enroll 200 adults with active pulmonary tuberculosis (TB; among whom 40 have HIV co-infections) at the time of TB diagnosis in S India. The intervention will include daily vitamin D supplementation in 3 treatment arms (600, 2000, and 4000 IU vitamin D), compared to placebo, for 12 months. The investigators' primary objectives are to assess how vitamin D supplementation affects immunity (immunological markers, immune competence) and serum vitamin D levels. Secondary outcomes include TB treatment outcomes (successful sputum smear conversion, relapse) in all patients, and human immunodeficiency virus (HIV) disease progression among a subset of patients with HIV co-infection.

ELIGIBILITY:
Inclusion Criteria:

* Active TB diagnosis by GeneXpert
* HIV infection status (according to AMC HIV clinic medical records of enzyme-linked immunosorbent assay [ELISA] results)

Exclusion Criteria:

* Children (<18 years of age)
* 60 years of age
* Pregnant at baseline
* Other severe complications or illnesses requiring hospitalization
* Received TB treatment for greater than 4 weeks in the past 5 years
* Refused to participate
* Residing in a geographic location > 1 hour from AMC (by public transit)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-06 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Immune function | One year
  Immune responses will be assessed by the superoxide bursts and proteolytic capacities of macrophages and monocytes. Activity indexes will be assessed by comparing mean substrate and calibration fluorescence.
Cell-mediated immunological markers | One year
  T cells
Vitamin D status | One year
  Serum 25(OH)D concentrations

SECONDARY OUTCOMES:
TB treatment outcomes | One year
  TB treatment success and relapse
HIV disease progression | One year
  WHO HIV disease stages

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Mehta, MBBS, ScD, Principal Investigator — Cornell University (U.S.); Wesley Bonam, BSc, MBBS, FAIMS, MRSH, Principal Investigator — Arogyavaram Medical Centre (India)
Locations (2):
- Cornell University, Ithaca, New York, United States
- Arogyavaram Medical Centre (AMC), Madanapalle, India